CLINICAL TRIAL: NCT02229825
Title: An Eight-week, Randomized, Double-blind, Two Parallel Groups, Study to Assess Clinical Response of Duloxetine 60 mg and 120 mg Per Day in Patients Hospitalized for Severe Depression
Brief Title: Study to Assess Clinical Response of Duloxetine in Patients Hospitalized for Severe Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1208.24
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Duloxetine 60 mg (Experimental): Duloxetine 60 mg
  Interventions: Drug: Duloxetine; Drug: Placebo
- Duloxetine 120 mg (Experimental): Duloxetine 120 mg
  Interventions: Drug: Duloxetine; Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Capsule
Drug: Placebo — Capsule

SUMMARY:
Study to assess efficacy of Duloxetine 120 mg and Duloxetine 60 mg in patients hospitalized for severe depression after 4 weeks of treatment. To evaluate the rescue option in non-responding patients. Safety of Duloxetine will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of 18 years of age at the screening visit or older
2. Meet criteria for severe Major Depressive Disorder (MDD)
3. Montgomery-Asberg-depression rating scale (MADRS) total score ≥ 30 and the 6-item Hamilton Depression scale (HAMD-6) score ≥12 at both screening (V1) visit and baseline (V2) visits
4. Clinical Global Impression of Severity (CGI-Severity) score ≥4 at both screening visit and baseline visit.
5. Requirement of hospitalization (not for social or other non-medical reasons) at screening visit and at least up to Visit 4
6. Patient willing and able to comply with the requirement for hospitalization and with all scheduled visits, tests and procedures required by the protocol
7. Have a level of understanding sufficient to provide informed consent and to communicate with the investigators and site personnel. Informed consent document must be signed at screening visit, in accordance with Good Clinical Practice (GCP) and local regulatory requirements, prior to any study procedure

Exclusion Criteria:

1. More than two previous episodes of major depression that did not respond to adequate doses and duration (minimum of 6 weeks) of two different antidepressant therapies
2. Lack of response to at least two antidepressant therapies given at adequate doses for at least 6 weeks for the current depressive episode
3. Concurrent presence of symptoms fulfilling criteria for any Axis I disorder other than anxiety disorders (with exception of the Obsessive-Compulsive Disorder (OCD)) or Major Depressive Disorder, in the investigator's judgment
4. Any previous diagnosis of a bipolar disorder, schizophrenia or OCD
5. Depression with catatonic features, depression with post-partum onset, or organic mental disorders
6. The presence of an Axis II disorder
7. MDD with psychotic features requiring neuroleptic treatment and/or interfering with patient's ability to provide informed consent, at investigator's discretion
8. History of substance abuse or dependence within the past year, excluding nicotine and caffeine, but including alcohol or benzodiazepines
9. Positive urine screen for drug abuse (cannabinoids, cocaine, opiates including methadone, or amphetamines) at screening
10. Epilepsy or a history of seizure disorder or of a treatment with anticonvulsant medication for epilepsy or seizures
11. Patients with acute liver injury (such as hepatitis) or severe cirrhosis (such as Child-Pugh Class C)
12. Known diagnosis of congenital galactosaemia, glucose or galactose malabsorption syndrome, or lactose deficiency
13. Patient with a known diagnosis of raised intraocular pressure, or at known risk of acute narrow-angle glaucoma
14. Serious medical illness or clinically significant laboratory abnormalities that, in the judgment of the investigator, are likely to require intervention/exclusion of study medication during the course of the study: cardiovascular (e.g. uncontrolled hypertension, abnormal initial ECG findings according to investigator judgement), respiratory, haematological, hepatic or gastrointestinal
15. End stage renal disease (estimated creatinine clearance ≤30 mL/min) and undergoing dialysis
16. Abnormal thyroid-stimulating hormone (TSH) concentrations, based on the performing laboratory's reference ranges. Patients must be clinically and chemically euthyroid at the time of randomization. Patients may be taking thyroid replacement therapy provided their dose is stable and their compliance is good for at least three months before the screening visit
17. Pregnancy (to be excluded by urine pregnancy test at screening visit) or breast-feeding
18. Sexually active woman of childbearing potential (i.e. not 6 months post-menopausal, or not surgically sterilized) not using a medically approved method of birth control (i.e. oral contraceptives, intrauterine device, or double-barrier) for at least one month prior to the screening visit and throughout the study
19. Participation in another clinical trial within 30 days prior to screening visit
20. Current treatment with Duloxetine for any indication and previous treatment with Duloxetine for psychiatric indications
21. Known hypersensitivity to Duloxetine or any of the inactive ingredients
22. History of oversensitivity to psychotropic drugs, in the investigator's judgment
23. Electro-convulsive Therapy (ECT) or Transcranial Magnetic Stimulation (TMS) within one year prior to screening visit and during the study
24. Initiation or discontinuation of depression-oriented psychotherapeutic treatment (e.g. behaviour therapy, psychoanalytic therapy, cognitive therapy, etc) within 6 weeks prior to screening visit, or planned use of such treatment at any time during the study
25. Treatment with a Monoamine Oxidase Inhibitor (MAOI) within 14 days prior to baseline visit or the potential need to use an MAOI during the study or within 5 days after discontinuation of duloxetine
26. Treatment with Fluoxetine within 30 days prior to baseline visit
27. Treatment with any excluded medication listed in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2007-02-09 (Actual); Primary Completion 2008-08-26 (Actual); Study Completion 2008-08-26 (Actual)

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized (1:1), double-blind, two parallel-group trial comparing the clinical response to duloxetine 60 milligram (mg) and 120 mg per day in patients hospitalized for severe depression over a 8-week treatment period. At Week 4, participants classified by the investigator as non-responders were up-titrated to receive the higher dose duloxetine.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 60 mg Duloxetine: 1 capsule of 60 milligram (mg) duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food for the first 4 weeks of treatment. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MADRS) as responders or non-responders. From week 4 to end of treatment responders (defined as ≥50% change in total MADRS score from baseline) continued with the same dosing regimen. Non-responders were up-titrated to 120 mg of duloxetine (1 capsule of 60 mg duloxetine in the morning and 1 capsule of 60 mg duloxetine + 1 placebo capsule in the evening).
- 120 mg Duloxetine: From day 1 to day 3, 1 capsule of 60 mg duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food. From day 4 until Visit 6, the dose was escalated to 120 mg (forced titration), with 1 capsule of duloxetine administered orally once daily in the morning and one in the evening. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MARDS) as responders or non-responders. From week 4 to end of treatment responders (defined as ≥50% change in total MADRS score from baseline) continued with the same dosing regimen. Non-responders were up-titrated to 3 capsules a day, remaining at 120 mg dose of duloxetine (1 capsule of 60 mg duloxetine in the morning and one in the evening and 1 placebo capsule in the evening).
Period: Overall Study
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Started | 167 | 172
Treated | 167 | 171
Completed | 143 | 142
Not Completed | 24 | 30
Not completed — Personal Reasons | 0 | 1
Not completed — Refused continuing medication | 7 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Lack of Efficacy | 4 | 10
Not completed — Adverse Event | 11 | 9
Not completed — Not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TRS): All randomised patients treated with at least one dose of duloxetine. Participants randomised but not treated with at least one dose of duloxetine were excluded, as they cannot contribute information on the drug effect.
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine | Total
Number analyzed (Participants) | 167 | 171 | 338
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (13.9) | 43.9 (12.7) | 44.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 38 | 87
  Male | 118 | 133 | 251
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 161 | 163 | 324
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Investigator Country [Count of Participants; unit: Participants]
  France | 64 | 64 | 128
  Italy | 7 | 6 | 13
  Russia | 81 | 84 | 165
  South Africa | 15 | 17 | 32
Montgomery-Asberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: score on scale] — The MADRS total score is used to measure the severity of depression. It is based on 10 items ranging from 0 to 6 each. The total score is calculated as the sum over the 10 items, ranging from 0 to 60. A lower score indicates a better outcome.
  Missing items (≤2 items) were replaced by the mean score of the participant's treatment group per time point. Otherwise, the MADRS total score was set to missing. Values are measured at baseline. TRS.
  score on scale | 36.1 (4.0) | 36.0 (4.6) | 36.1 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline to Week 4
Description: The MADRS total score is used to measure the severity of depression. It is based on 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts) scored from 0 to 6 each. The total score is calculated as the sum over the 10 items, ranging from 0 to 60. A lower score indicates a better outcome.
  Missing items (≤2 items) were replaced by the mean score of the participant's treatment group per time point. Otherwise, the MADRS total score was set to missing.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At baseline and at Week 4.
Population: Full Analysis Set (FAS): All participants who received at least one dose of duloxetine and who had at least one baseline value and one post-baseline value available for efficacy evaluation. Treatment regimen.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Units on a scale | -20.1 (10.6) | -19.9 (10.0)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs 120 mg Duloxetine; The null hypothesis was that the mean change in MADRS total score between week 4 and baseline was the same for the 2 duloxetine treatment groups; Test type: Other; p = 0.88, ANCOVA — p-value for treatment effect; ANCOVA with stratification factors (country and pretreatment) and baseline score and treatment as the main factor

2. Secondary Outcome: Change in Hamilton Depression 6-item Scale (HAMD-6) Total Score From Baseline to Week 1, 2, 3 and Week 4
Description: HAMD-6 is a 6-item rating instrument that assesses items thought to represent 'core' symptoms of depression. It was derived from standard 17-item Hamilton Depression Scale (HAMD-17) with assessment being restricted to items 1, 2, 7, 8, 10 and 13. The HAMD-6 score is calculated as the sum over the 6 items, ranging from 0 to 22, with a lower score indicating a better patient status.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At baseline and at Week 1, 2, 3 and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Units on a scale
  Change from baseline to week 1 | -3.1 (3.6) | -2.7 (3.3)
  Change from baseline to week 2 | -5.8 (4.6) | -5.2 (4.2)
  Change from baseline to week 3 | -7.2 (4.4) | -6.8 (4.4)
  Change from baseline to week 4 | -8.0 (4.8) | -8.1 (4.7)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs 120 mg Duloxetine; Comparison between treatment regimes at Week 4; Test type: Other; p = 0.86, ANCOVA — Treatment effect; Analysis of covariance (ANCOVA) with stratification factors and HAMD6 baseline as covariates and treatment regimen as main factor

3. Secondary Outcome: Change in Hamilton Depression 6-item Scale (HAMD-6) Total Score From Baseline to Week 6 and Week 8 - by Post-week 4 Treatment Groups
Description: HAMD-6 is a 6-item rating instrument that assesses items thought to represent 'core' symptoms of depression. It was derived from standard 17-item Hamilton Depression Scale (HAMD-17) with assessment being restricted to items 1, 2, 7, 8, 10 and 13. The HAMD-6 score is calculated as the sum over the 6 items, ranging from 0 to 22, with a lower score indicating a better patient status.
  Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At baseline and at Week 6 and Week 8.
Population: Full Analysis Set (FAS): All participants who received at least one dose of duloxetine and who had at least one baseline value and one post-baseline value available for efficacy evaluation. Only participants with non-missing values are reported. Post-week 4 treatment groups.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- 60 mg Duloxetine - Responder: 1 capsule of 60 milligram (mg) duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food for the first 4 weeks of treatment. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MADRS) as responders or non-responders. From week 4 to end of treatment responders (defined as ≥50% change in total MADRS score from baseline) continued with the same dosing regimen.
- 60 mg Duloxetine - Non-Responder: 1 capsule of 60 milligram (mg) duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food for the first 4 weeks of treatment. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MADRS) as responders or non-responders. From week 4 to end of treatment, non-responders were up-titrated to 120 mg of duloxetine (1 capsule of 60 mg duloxetine in the morning and 1 capsule of 60 mg duloxetine + 1 placebo capsule in the evening).
- 120 mg Duloxetine - Responder: From day 1 to day 3, 1 capsule of 60 mg duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food. From day 4 until Visit 6, the dose was escalated to 120 mg (forced titration), with 1 capsule of duloxetine administered orally once daily in the morning and one in the evening. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MARDS) as responders or non-responders. From week 4 to end of treatment, responders (defined as ≥50% change in total MADRS score from baseline) continued with the same dosing regimen.
- 120 mg Duloxetine - Non-Responder: From day 1 to day 3, 1 capsule of 60 mg duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food. From day 4 until Visit 6, the dose was escalated to 120 mg (forced titration), with 1 capsule of duloxetine administered orally once daily in the morning and one in the evening. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MARDS) as responders or non-responders. From week 4 to end of treatment, non-responders were up-titrated to 3 capsules a day, remaining at 120 mg dose of duloxetine (1 capsule of 60 mg duloxetine in the morning and one in the evening and 1 placebo capsule in the evening).
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-Responder | 120 mg Duloxetine - Responder | 120 mg Duloxetine - Non-Responder
Number analyzed (Participants) | 96 | 70 | 106 | 64
Units on a scale
  Change from baseline to week 6: number analyzed (Participants) | 96 | 55 | 106 | 48
  Change from baseline to week 6 | -11.6 (3.5) | -6.4 (4.4) | -11.8 (3.3) | -5.5 (4.4)
  Change from baseline to week 8 | -12.3 (3.4) | -7.6 (5.1) | -12.5 (3.0) | -6.7 (5.4)
Statistical Analysis 1: Comparison: 60 mg Duloxetine - Responder; Within-group comparisons, week 8 versus baseline; Test type: Other; p < 0.0001, Signed Rank test
Statistical Analysis 2: Comparison: 60 mg Duloxetine - Non-Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p < 0.0001, Singed Rank test
Statistical Analysis 3: Comparison: 120 mg Duloxetine - Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p < 0.0001, Singed Rank test
Statistical Analysis 4: Comparison: 120 mg Duloxetine - Non-Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p < 0.0001, Signed Rank test

4. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline to Week 1, 2 and Week 3
Description: The MADRS total score is used to measure the severity of depression. It is based total score is based on 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts) ranging from 0 to 6 each. The total score is calculated as the sum over the 10 items, ranging from 0 to 60. A lower score indicates a better outcome.
  Missing items (≤2 items) were replaced by the mean score of the participant's treatment group per time point. Otherwise, the MADRS total score was set to missing.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At baseline and at Week 1, 2 and Week 3.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Units on a scale
  Change from baseline to Week 1 | -8.3 (8.0) | -7.6 (7.3)
  Change from baseline to Week 2 | -14.7 (9.9) | -13.5 (8.9)
  Change from baseline to Week 3 | -18.1 (9.8) | -16.9 (9.3)

5. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline to Week 6 and Week 8 - by Post-week 4 Treatment Groups
Description: The MADRS total score is based on 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts) ranging from 0 to 6 each. The total score is calculated as the sum over the 10 items, ranging from 0 to 60. A lower score indicates a better outcome.
  Missing items (≤2 items) were replaced by the mean score of the participant's treatment group per time point. Otherwise, the MADRS total score was set to missing.
  Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At baseline and at Week 6 and Week 8.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- 60 mg Duloxetine - Responder: 1 capsule of 60 milligram (mg) duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food for the first 4 weeks of treatment. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MADRS) as responders or non-responders. From week 4 to end of treatment, responders (defined as ≥50% change in total MADRS score from baseline) continued with the same dosing regimen.
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-responder | 120 mg Duloxetine - Responder | 120 mg Duloxetine - Non-responder
Number analyzed (Participants) | 96 | 70 | 106 | 64
Units on a scale
  Change from baseline to week 6: number analyzed (Participants) | 96 | 55 | 106 | 48
  Change from baseline to week 6 | -28.3 (7.9) | -16.1 (9.4) | -28.1 (6.6) | -14.8 (10.4)
  Change from baseline to week 8 | -29.8 (7.3) | -19.0 (11.8) | -29.5 (6.6) | -17.2 (12.3)
Statistical Analysis 1: Comparison: 60 mg Duloxetine - Responder; Within group comparisons were performed at week 8 versus baseline; Test type: Other; p < 0.0001, McNemar
Statistical Analysis 2: Comparison: 60 mg Duloxetine - Non-responder; Within group comparisons were performed at week 8 versus baseline; Test type: Other; p < 0.0001, McNemar
Statistical Analysis 3: Comparison: 120 mg Duloxetine - Responder; Within group comparisons were performed at week 8 versus baseline; Test type: Other; p < 0.0001, McNemar
Statistical Analysis 4: Comparison: 120 mg Duloxetine - Non-responder; Within group comparisons were performed at week 8 versus baseline; Test type: Other; p < 0.0001, McNemar

6. Secondary Outcome: Percentage of Responders at Week 1, 2, 3 and Week 4 According to Montgomery-Asberg Depression Rating Scale (MADRS) Scale
Description: Percentage of patient 'responders', i.e. patients with at least a 50% improvement in MADRS scores from baseline.
  The MADRS total score is used to measure the severity of depression. It is based on 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts) ranging from 0 to 6 each. The total score is calculated as the sum over the 10 items, ranging from 0 to 60. A lower score indicates a better outcome.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At week 1, 2, 3 and week 4.
Population: Full Analysis Set (FAS): All participants who received at least one dose of duloxetine and who had at least one baseline value and one post-baseline value available for efficacy evaluation. Treatment-regimen.
Measure: Number; unit: Percentage of Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Percentage of Participants
  Week 1 | 14.5 | 8.2
  Week 2 | 33.7 | 31.2
  Week 3 | 50.0 | 46.5
  Week 4 | 59.0 | 64.1
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs 120 mg Duloxetine; Treatment groups were compared regarding the number of responders and non-responders at week 4, using a logistic regression with stratification factors (country and pretreatment) and baseline scores as covariates and treatment regimen as main factor; Test type: Other; p = 0.32, Regression, Logistic — Treatment effect

7. Secondary Outcome: Percentage of Responders at Week 6 and Week 8 According to Montgomery-Asberg Depression Rating Scale (MADRS) Scale - by Post-week 4 Treatment Groups
Description: Percentage of patient 'responders', i.e. patients with at least a 50% improvement in MADRS scores from baseline.
  The MADRS total score is used to measure the severity of depression. It is based on 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts) ranging from 0 to 6 each. The total score is calculated as the sum over the 10 items, ranging from 0 to 60. A lower score indicates a better outcome.
  Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At week 6 and week 8.
Population: Full Analysis Set (FAS): All participants who received at least one dose of duloxetine and who had at least one baseline value and one post-baseline value available for efficacy evaluation. Post-week 4 treatment groups.
Measure: Number; unit: Percentage of Participants
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-Responder | 120 mg Duloxetine - Responder | 120 mg Duloxetine - Non-Responder
Number analyzed (Participants) | 96 | 70 | 106 | 64
Percentage of Participants
  Week 6 | 94.8 | 52.9 | 98.1 | 39.1
  Week 8 | 93.8 | 65.7 | 98.1 | 54.7

8. Secondary Outcome: Percentage of Responders at Week 1, 2, 3 and Week 4 According to Hamilton Depression 6-item Scale (HAMD-6)
Description: Percentage of patient 'responders', i.e. patients with at least a 50% improvement in HAMD-6 scores from baseline.
  HAMD-6 is a 6-item rating instrument that assesses items thought to represent 'core' symptoms of depression. It was derived from standard 17-item Hamilton Depression Scale (HAMD-17) with assessment being restricted to items 1, 2, 7, 8, 10 and 13. The HAMD-6 score is calculated as the sum over the 6 items, ranging from 0 to 22, with a lower score indicating a better patient status.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At week 1, 2, 3 and week 4.
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Percentage of Participants
  Week 1 | 12.0 | 10.0
  Week 2 | 32.5 | 26.5
  Week 3 | 42.8 | 44.1
  Week 4 | 55.4 | 58.2
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs 120 mg Duloxetine; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.57, Regression, Logistic — Treatment effect

9. Secondary Outcome: Percentage of Responders at Week 6 and Week 8 According to Hamilton Depression 6-item Scale (HAMD-6) - by Post-week 4 Treatment Group
Description: Percentage of patient 'responders', i.e. patients with at least a 50% improvement in HAMD-6 scores from baseline.
  HAMD-6 is a 6-item rating instrument that assesses items thought to represent 'core' symptoms of depression. It was derived from standard 17-item Hamilton Depression Scale (HAMD-17) with assessment being restricted to items 1, 2, 7, 8, 10 and 13. The HAMD-6 score is calculated as the sum over the 6 items, ranging from 0 to 22, with a lower score indicating a better patient status.
  Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At week 6 and week 8.
Population: Full-Analysis Set (FAS): This included all participants who received at least one dose of duloxetine and who had at least one baseline value and one post-baseline value available for efficacy evaluation. Post-week 4 treatment groups.
Measure: Number; unit: Percentage of participants
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-Responder | 120 mg Duloxetine - Responder | 120 mg Duloxetine - Non-Responder
Number analyzed (Participants) | 96 | 70 | 106 | 64
Percentage of participants
  Week 6 | 90.6 | 47.1 | 90.6 | 31.3
  Week 8 | 92.7 | 60.0 | 95.3 | 46.9

10. Secondary Outcome: Percentage of Patients Reaching Remission at Week 8
Description: Remission is defined as a total Montgomery-Asberg Depression Rating Scale (MADRS) score of ≤ 12 at week 8.
  The MADRS total score is based on 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts) ranging from 0 to 6 each and a total MADRS score ranging from 0 to 60.
  Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At week 8.
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-Responder | 120 mg Duloxetine - Responder | 120 mg Duloxetine - Non-Responder
Number analyzed (Participants) | 96 | 70 | 106 | 64
Percentage of participants
  No | 11.5 | 58.6 | 11.3 | 71.9
  Yes | 88.5 | 41.4 | 88.7 | 28.1

11. Secondary Outcome: Clinical Global Impressions Scales of Severity of Illness (CGI-SI): Number of Patients Per Score at Baseline, Week 1, 2, 3 and Week 4
Description: Clinical Global Impression (CGI) scales were developed as an independent, simple way for clinicians to make overall evaluations of a patient's disease status. The CGI-SI assess the severity of illness, with the following question: "Considering your total clinical experience with the particular population, how mentally ill is the patient at this time?". The CGI-SI ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). A higher score indicates a worse patient status.
  Reported is the number of patients per score by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
  At week 4 treatment groups were compared using the Cochran Mantel-Haenszel test with stratification by centre.
Time Frame: At baseline and at week 1, 2, 3 and week 4.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Participants
  Baseline: Not at all ill | 0 | 0
  Baseline: Borderline ill | 0 | 0
  Baseline: Mildly ill | 0 | 0
  Baseline: Moderately ill | 33 | 30
  Baseline: Markedly ill | 93 | 87
  Baseline: Severely ill | 40 | 51
  Baseline: Most extremely ill | 0 | 2
  Week 1: Not at all ill | 0 | 1
  Week 1: Borderline ill | 6 | 3
  Week 1: Mildly ill | 20 | 17
  Week 1: Moderately ill | 62 | 64
  Week 1: Markedly ill | 62 | 68
  Week 1: Severely ill | 16 | 17
  Week 1: Most extremely ill | 0 | 0
  Week 2: Not at all ill | 8 | 6
  Week 2: Borderline ill | 22 | 11
  Week 2: Mildly ill | 45 | 48
  Week 2: Moderately ill | 53 | 61
  Week 2: Markedly ill | 33 | 39
  Week 2: Severely ill | 5 | 5
  Week 2: Most extremely ill | 0 | 0
  Week 3: Not at all ill | 17 | 9
  Week 3: Borderline ill | 30 | 29
  Week 3: Mildly ill | 48 | 56
  Week 3: Moderately ill | 41 | 49
  Week 3: Markedly ill | 27 | 22
  Week 3: Severely ill | 3 | 4
  Week 3: Most extremely ill | 0 | 1
  Week 4: Not at all ill | 28 | 17
  Week 4: Borderline ill | 35 | 46
  Week 4: Mildly ill | 34 | 50
  Week 4: Moderately ill | 47 | 33
  Week 4: Markedly ill | 18 | 17
  Week 4: Severely ill | 3 | 6
  Week 4: Most extremely ill | 1 | 1
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs 120 mg Duloxetine; At week 4 CGI-S items were pooled to reduce the possible number of classes before formal testing. The 3 classes used (instead of 7 items) were: 1-2: "normal", 3-5: "moderate", 6-7: "severe. Treatment groups were compared using the Cochran Mantel-Haenszel test with stratification by centre; Test type: Other; p = 0.68, Cochran-Mantel-Haenszel; Stratified by country, 60 mg vs. 120 mg

12. Secondary Outcome: Clinical Global Impressions Scales of Severity of Illness (CGI-SI): Number of Patients Per Score at Week 6 and Week 8 - by Post-week 4 Treatment Groups
Description: The Clinical Global Impressions scales of Severity of Illness (CGI-SI) were developed as an independent, simple way for clinicians to make overall evaluations of a patient's disease status. The CGI-SI assess the severity of illness, with the following question: "Considering your total clinical experience with the particular population, how mentally ill is the patient at this time?".
  The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). A higher score indicates a worse patient status.
  Number of patients per score is reported. Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
  At week 8, within-group comparison versus week 4 was performed for each post-week 4 treatment group using Mc Nemar test.
Time Frame: At week 6 and week 8.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- 60 mg Duloextine - Non-Responder: 1 capsule of 60 milligram (mg) duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food for the first 4 weeks of treatment. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MADRS) as responders or non-responders. From week 4 to end of treatment, non-responders were up-titrated to 120 mg of duloxetine (1 capsule of 60 mg duloxetine in the morning and 1 capsule of 60 mg duloxetine + 1 placebo capsule in the evening).
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloextine - Non-Responder | 120 mg Duloxetine - Responder | 120 mg Duloxetine - Non-Responder
Number analyzed (Participants) | 96 | 70 | 106 | 64
Participants
  Week 6: Not at all ill | 38 | 1 | 41 | 2
  Week 6: Borderline ill | 31 | 9 | 40 | 6
  Week 6: Mildly ill | 21 | 32 | 21 | 16
  Week 6: Moderately ill | 4 | 11 | 3 | 19
  Week 6: Markedly ill | 1 | 12 | 1 | 14
  Week 6: Severely ill | 1 | 4 | 0 | 6
  Week 6: Most extremely ill | 0 | 1 | 0 | 1
  Week 8: Not at all ill | 51 | 6 | 54 | 5
  Week 8: Borderline ill | 30 | 23 | 39 | 13
  Week 8: Mildly ill | 10 | 19 | 10 | 15
  Week 8: Moderately ill | 4 | 6 | 2 | 11
  Week 8: Markedly ill | 1 | 10 | 1 | 12
  Week 8: Severely ill | 0 | 5 | 0 | 7
  Week 8: Most extremely ill | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: 60 mg Duloxetine - Responder; At week 8, within-group comparison versus week 4 was performed; Test type: Other; p < 0.0001, Signed Rank test; Statistic = -528 — Difference is value at week 8 minus week 4
Statistical Analysis 2: Comparison: 60 mg Duloextine - Non-Responder; At week 8, within-group comparison versus week 4 was performed; Test type: Other; p < 0.0001, Signed Rank test; Statistic = -540 — Difference is value at week 8 minus week 4
Statistical Analysis 3: Comparison: 120 mg Duloxetine - Responder; At week 8, within-group comparison versus week 4 was performed; Test type: Other; p < 0.0001, Signed Rank test; Statistic = -1024.5 — Difference is value at week 8 minus week 4
Statistical Analysis 4: Comparison: 120 mg Duloxetine - Non-Responder; At week 8, within-group comparison versus week 4 was performed; Test type: Other; p < 0.0001, Signed Rank test; Statistic = -279 — Difference is value at week 8 minus week 4

13. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Scale: Number of Patients Per Score at Week 1, 2, 3 and Week 4
Description: The Clinical Global Impression of Improvement (CGI-I) scale was developed as an independent, simple way for clinicians to make overall evaluations of a patients disease status. The CGI-I rates the total improvement with the following question:
  "Compared to the patients condition at admission, how much has he or she changed?". The scale ranges from 1 (very much improved) to 7 (very much worse). A higher score indicates a worse patient status.
  Number of patients per score is reported. Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
  At week 4 treatment groups were compared using the Cochran Mantel-Haenszel test with stratification by centre.
Time Frame: At week 1, 2, 3 and week 4.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Participants
  Week 1: Very much improved | 5 | 2
  Week 1: Much improved | 29 | 25
  Week 1: Minimally improved | 75 | 84
  Week 1: No change | 52 | 55
  Week 1: Minimally worse | 5 | 4
  Week 1: Much worse | 0 | 0
  Week 1: Very much worse | 0 | 0
  Week 2: Very much improved | 22 | 16
  Week 2: Much improved | 64 | 60
  Week 2: Minimally improved | 61 | 76
  Week 2: No change | 13 | 17
  Week 2: Minimally worse | 5 | 1
  Week 2: Much worse | 1 | 0
  Week 2: Very much worse | 0 | 0
  Week 3: Very much improved | 31 | 25
  Week 3: Much improved | 76 | 78
  Week 3: Minimally improved | 46 | 53
  Week 3: No change | 8 | 11
  Week 3: Minimally worse | 4 | 3
  Week 3: Much worse | 1 | 0
  Week 3: Very much worse | 0 | 0
  Week 4: Very much improved | 38 | 44
  Week 4: Much improved | 67 | 78
  Week 4: Minimally improved | 45 | 34
  Week 4: No change | 10 | 11
  Week 4: Minimally worse | 3 | 2
  Week 4: Much worse | 2 | 1
  Week 4: Very much worse | 1 | 0
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs 120 mg Duloxetine; [analysis description as in outcome 11, analysis 1]; Test type: Other — No formal hypothesis was tested; p = 0.07, Cochran-Mantel-Haenszel — Stratified by country, 60 mg vs. 120 mg

14. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Scale: Number of Patients Per Score at Week 6 and Week 8 - by Post-week 4 Treatment Groups
Description: Clinical Global Impression (CGI) scale was developed as an independent, simple way for clinicians to make overall evaluations of a patients disease status. The CGI-I rates the total improvement with the following question:
  "Compared to the patients condition as admission, how much has he or she changed?". The CGI-I score ranges from 1 (very much improved) to 7 (very much worse). A higher score indicates a worse patient outcome.
  Number of patients per score is reported. Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At week 6 and week 8.
Population: Full Analysis Set (FAS): All participants who received at least one dose of duloxetine and who had at least one baseline value and one post-baseline value available for efficacy evaluation. Post-week 4 treatment group.
Measure: Count of Participants; unit: Participants
Groups:
- 120 mg Duloxeting - Non-Responder: From day 1 to day 3, 1 capsule of 60 mg duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food. From day 4 until Visit 6, the dose was escalated to 120 mg (forced titration), with 1 capsule of duloxetine administered orally once daily in the morning and one in the evening. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MARDS) as responders or non-responders. From week 4 to end of treatment, non-responders were up-titrated to 3 capsules a day, remaining at 120 mg dose of duloxetine (1 capsule of 60 mg duloxetine in the morning and one in the evening and 1 placebo capsule in the evening).
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-Responder | 120 mg Duloxetine - Responder | 120 mg Duloxeting - Non-Responder
Number analyzed (Participants) | 96 | 70 | 106 | 64
Participants
  Week 6: Very much improved | 55 | 6 | 61 | 6
  Week 6: Much improved | 35 | 39 | 38 | 27
  Week 6: Minimally improved | 3 | 12 | 5 | 15
  Week 6: No change | 3 | 6 | 2 | 13
  Week 6: Minimally worse | 0 | 3 | 0 | 1
  Week 6: Much worse | 0 | 3 | 0 | 2
  Week 6: Very much worse | 0 | 1 | 0 | 0
  Week 8: Very much improved | 64 | 12 | 71 | 8
  Week 8: Much improved | 25 | 36 | 30 | 26
  Week 8: Minimally improved | 5 | 7 | 2 | 13
  Week 8: No change | 2 | 7 | 2 | 14
  Week 8: Minimally worse | 0 | 4 | 1 | 1
  Week 8: Much worse | 0 | 3 | 0 | 2
  Week 8: Very much worse | 0 | 1 | 0 | 0

15. Secondary Outcome: Patient Global Impressions of Improvement (PGI-I) Score: Number of Patients Per Score at Week 1, 2, 3 and Week 4
Description: Patient Global Impression of Improvement scale is a patient-rated instrument that measures the improvement of the patient's symptoms, ranging from 1 (very much better) to 7 (much worse). A higher score indicates a worse outcome.
  Number of patients per score is reported. Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
  At week 4 treatment groups were compared using the Cochran Mantel-Haenszel test with stratification by centre.
Time Frame: At week 1, 2, 3 and week 4.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Participants
  Week 1: Missing | 2 | 0
  Week 1: Very much better | 7 | 7
  Week 1: Much better | 45 | 26
  Week 1: A little better | 62 | 83
  Week 1: No change | 40 | 47
  Week 1: A little worse | 8 | 7
  Week 1: Much worse | 1 | 0
  Week 1: Very much worse | 1 | 0
  Week 2: Missing | 2 | 0
  Week 2: Very much better | 22 | 20
  Week 2: Much better | 63 | 56
  Week 2: A little better | 56 | 73
  Week 2: No change | 17 | 18
  Week 2: A little worse | 3 | 2
  Week 2: Much worse | 1 | 1
  Week 2: Very much worse | 2 | 0
  Week 3: Missing | 1 | 0
  Week 3: Very much better | 35 | 34
  Week 3: Much better | 66 | 62
  Week 3: A little better | 49 | 50
  Week 3: No change | 10 | 19
  Week 3: A little worse | 3 | 2
  Week 3: Much worse | 0 | 2
  Week 3: Very much worse | 2 | 1
  Week 4: Missing | 1 | 0
  Week 4: Very much better | 43 | 49
  Week 4: Much better | 66 | 64
  Week 4: A little better | 38 | 37
  Week 4: No change | 11 | 12
  Week 4: A little worse | 3 | 3
  Week 4: Much worse | 0 | 4
  Week 4: Very much worse | 4 | 1
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs 120 mg Duloxetine; Before testing, PGI-I items were pooled to reduce the possible number of classes. The 3 classes used (instead of 7 items) were: 1-2= "improved", 3-5="Stable", 6-7="Worsened". At week 4 treatment groups were compared using the Cochran Mantel-Haenszel test with stratification by centre; Test type: Other; p = 1.00, Cochran-Mantel-Haenszel; CMH statistic = 0.00

16. Secondary Outcome: Patient Global Impressions of Improvement (PGI-I) Score: Number of Patients Per Score at Week 6 and Week 8 - by Post-week 4 Treatment Groups
Description: Patient Global Impression of Improvement scale is a patient-rated instrument that measures the improvement of the patient's symptoms, ranging from 1 (very much better) to 7 (much worse). A higher score indicates a worse outcome.
  Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At week 6 and week 8.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- 120mg Duloxetine - Responder: From day 1 to day 3, 1 capsule of 60 mg duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food. From day 4 until Visit 6, the dose was escalated to 120 mg (forced titration), with 1 capsule of duloxetine administered orally once daily in the morning and one in the evening. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MARDS) as responders or non-responders. From week 4 to end of treatment, responders (defined as ≥50% change in total MADRS score from baseline) continued with the same dosing regimen.
- 120mg Duloxetine - Non-Responder: From day 1 to day 3, 1 capsule of 60 mg duloxetine was administered orally once daily in the morning and 1 capsule of placebo was administered orally once daily in the evening, each with a glass of water, with or without food. From day 4 until Visit 6, the dose was escalated to 120 mg (forced titration), with 1 capsule of duloxetine administered orally once daily in the morning and one in the evening. At Visit 6 (week 4) patients were classified by the Montgomery-Asberg Depression Rating Scale (MARDS) as responders or non-responders. From week 4 to end of treatment, non-responders were up-titrated to 3 capsules a day, remaining at 120 mg dose of duloxetine (1 capsule of 60 mg duloxetine in the morning and one in the evening and 1 placebo capsule in the evening).
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-Responder | 120mg Duloxetine - Responder | 120mg Duloxetine - Non-Responder
Number analyzed (Participants) | 96 | 70 | 106 | 64
Participants
  Week 6: Missing | 0 | 1 | 0 | 0
  Week 6: Very much better | 48 | 7 | 61 | 5
  Week 6: Much better | 37 | 33 | 34 | 25
  Week 6: A little better | 5 | 17 | 7 | 18
  Week 6: No change | 4 | 5 | 4 | 12
  Week 6: A little worse | 1 | 2 | 0 | 1
  Week 6: Much worse | 1 | 1 | 0 | 2
  Week 6: Very much worse | 0 | 4 | 0 | 1
  Week 8: Missing | 0 | 1 | 0 | 0
  Week 8: Very much better | 62 | 17 | 72 | 17
  Week 8: Much better | 26 | 25 | 27 | 10
  Week 8: A little better | 4 | 11 | 4 | 18
  Week 8: No change | 4 | 8 | 2 | 15
  Week 8: A little worse | 0 | 2 | 1 | 1
  Week 8: Much worse | 0 | 2 | 0 | 2
  Week 8: Very much worse | 0 | 4 | 0 | 1

17. Secondary Outcome: Change in Hamilton Scale of Anxiety (HAMA) Score From Baseline to Week 4
Description: HAMA scale consists of 14 items to measure the severity of anxiety symptoms. Each item ranges from 0 (not present) to 4 (very severe). The total score is calculated as the sum over all items, ranging from 0 to 56, with a higher score implying a worse outcome. Change from baseline to week 4 is reported. Reduction in the score over time is interpreted as improvement in the patient´s status.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At baseline and at week 4.
Population: Only participants in the FAS and with non-missing values for this endpoint were included in the analysis. Treatment regimen.
Measure: Mean (Standard Deviation); unit: Units on a score
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 165 | 168
Units on a score | -13.0 (9.0) | -13.6 (9.0)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs 120 mg Duloxetine; Comparison between HAMA scores between treatment regimens; Test type: Other; p = 0.92, ANCOVA — Treatment effect

18. Secondary Outcome: Change in Hamilton Scale of Anxiety (HAMA) Score From Baseline to Week 8 - by Post-week 4 Treatment Groups
Description: HAMA scale consists of 14 items to measure the severity of anxiety symptoms. Each item ranges from 0 (not present) to 4 (very severe). The total score is calculated as the sum over all items, ranging from 0 to 56, with a higher score implying a worse outcome. Change from baseline to week 8 is reported. Reduction in the score over time is interpreted as improvement in the patient´s status.
  Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At baseline and at week 8.
Population: Only participants in the FAS and with non-missing values for this endpoint were included in the analysis. Post-week 4 treatment groups.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-Responder | 120 mg Duloxetine - Responder | 120 mg Duloxetine - Non-Responder
Number analyzed (Participants) | 96 | 69 | 106 | 62
Score on a scale | -19.6 (7.9) | -12.1 (10.1) | -21.0 (7.6) | -10.8 (10.0)
Statistical Analysis 1: Comparison: 60 mg Duloxetine - Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p < 0.0001, Student statistic t-test
Statistical Analysis 2: Comparison: 120 mg Duloxetine - Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p < 0.0001, Student statistic t-test
Statistical Analysis 3: Comparison: 60 mg Duloxetine - Non-Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p < 0.0001, Student statistic t-test
Statistical Analysis 4: Comparison: 120 mg Duloxetine - Non-Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p < 0.0001, Student statistic t-test

19. Secondary Outcome: Reason for Living (RFL) Questionaire at Baseline
Description: The Reason for Living (RFL) questionnaire is a self-report instrument, to evaluate a variety of expectations and adaptive beliefs for living, if suicide is considered.
  The RFL is thought to assess 6 domains of reasons for living: 1) survival and coping beliefs, 2) responsibility to family, 3) child related concerns, 4) fear of suicide, 5) fear of social disapproval, and 6) moral objections.
  The RFL uses a 6-point rating scale, with the total score ranging from 1 "not at all important" and to 6 "extremely important". A higher score indicates more reasons to live (i.e. better outcome).
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At baseline.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 162 | 167
Score on a scale | 3.8 (1.1) | 3.7 (1.0)

20. Secondary Outcome: Change From Baseline to Week 8 in Reason for Living (RFL) Questionnaire - by Post-week 4 Treatment Groups
Description: The Reason for Living (RFL) questionnaire is a self-report instrument, to evaluate a variety of expectations and adaptive beliefs for living, if suicide is considered.
  The RFL is thought to assess 6 domains of reasons for living: 1) survival and coping beliefs, 2) responsibility to family, 3) child related concerns, 4) fear of suicide, 5) fear of social disapproval, and 6) moral objections.
  The RFL uses a 6-point rating scale, with the total score ranging from 1 "not at all important" and to 6 "extremely important". A higher score indicates more reasons to live (i.e. better outcome).
  Results are reported by 'post-week 4 treatment groups' (treatment regimen (60 vs. 120 mg duloxetine) and responder/non-responder status). Patients were assigned their responder status at Visit 6 and the data were retrospectively divided into these groups.
Time Frame: At baseline and at week 8.
Population: Only participants included in the FAS and with non-missing values for this endpoint were included in the analysis. Post-week 4 treatment groups.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 60 mg Duloxetine - Responder | 60 mg Duloxetine - Non-Responder | 120 mg Duloxetine - Responder | 120 mg Duloxetine - Non-Responder
Number analyzed (Participants) | 93 | 59 | 100 | 57
Score on a scale | 0.7 (0.9) | 0.4 (0.8) | 0.8 (0.8) | 0.1 (0.9)
Statistical Analysis 1: Comparison: 60 mg Duloxetine - Responder; Within-group comparison, Week 8 versus baseline; Test type: Other; p < 0.0001, Student statistic t-test
Statistical Analysis 2: Comparison: 60 mg Duloxetine - Non-Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p = 0.001, Student statistic t-test
Statistical Analysis 3: Comparison: 120 mg Duloxetine - Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p < 0.0001, Student statistic t-test
Statistical Analysis 4: Comparison: 120 mg Duloxetine - Non-Responder; Within-group comparison, week 8 versus baseline; Test type: Other; p = 0.28, Student statistic t-test

21. Secondary Outcome: Number of Patients With Intake of Concomitant Medication for Anxiety and Sleep
Description: Number of patients with concomitant medication for anxiety and sleep taken at different timepoints.
  V1: Screening V2: Baseline V3: Week 1 V4: Week2 V5: Week 3 V6: Week 4 V7: Week 6 V8: Week 8.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: 1 week prior to baseline and at baseline, week 1, 2, 3, 4, 5, 6, 7, 8 and week 10.
Population: Only participants included in the treated set and with non-missing values for this endpoint were included in the analysis. Treatment regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 125 | 123
Participants
  Number of patients with medication taken before V1 | 65 | 59
  Number of patients with medication taken between V1 - V2 | 93 | 88
  Number of patients with medication taken between V2 - V3 | 95 | 89
  Patients with medication taken between V3 - V4 | 80 | 84
  Number of patients with medication taken between V4 - V5 | 62 | 67
  Number of patients with medication taken between V5 - V6 | 55 | 58
  Number of patients with medication taken between V6 - V7 | 47 | 49
  Number of patients with medication taken between V7 - V8 | 51 | 52
  Number of patients with medication taken after V8 (week 10) | 18 | 10
  Number of patients with medication not taken between two consecutive visits | 8 | 8

22. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Event
Description: Number of patients with any adverse event occuring during on-treatment phase.
  Results are reported for treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: From start of treatment until 3 days after end of treatment, up to 120 days.
Population: Treated Set (TRS): All randomised patients treated with at least one dose of duloxetine. Participants randomised but not treated with at least one dose of duloxetine were excluded, as they cannot contribute information on the drug effect. Treatment regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 167 | 171
Participants | 97 | 89

23. Secondary Outcome: Change From Baseline in Blood Pressure to Week 4 and Week 8
Description: Change from baseline in systolic and diastolic blood pressure (BP) to week 4 and week 8.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At baseline, at week 4 and week 8.
Population: Treated Set (TRS): All randomised patients treated with at least one dose of study medication. Patients randomised but not treated with at least one dose of study drug were excluded, as they cannot contribute information on the drug effect. Only patients with non-missing data for this endpoint were included.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 166 | 170
Millimeters of mercury (mmHg)
  Systolic BP: Change from baseline to week 4.: number analyzed (Participants) | 166 | 167
  Systolic BP: Change from baseline to week 4. | 2.0 (12.7) | 0.5 (13.2)
  Systolic BP: Change from baseline to week 8: number analyzed (Participants) | 163 | 168
  Systolic BP: Change from baseline to week 8 | 2.5 (13.0) | 2.0 (14.2)
  Diastolic BP: Change from baseline to week 4. | 1.9 (9.5) | 0.7 (9.6)
  Diastolic BP: Change from baseline to week 8 | 2.3 (9.6) | 2.5 (20.3)

24. Secondary Outcome: Change From Baseline in Weight to Week 4 and Week 8
Description: Change from baseline in weight to week 4 and week 8.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: At baseline, at week 4 and week 8.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 167 | 171
Kilogram (kg)
  Change from baseline to week 4: number analyzed (Participants) | 167 | 167
  Change from baseline to week 4 | 0.1 (2.0) | 0.0 (2.3)
  Change from baseline to week 8: number analyzed (Participants) | 163 | 168
  Change from baseline to week 8 | 0.5 (2.9) | 0.1 (2.8)

25. Secondary Outcome: Number of Patients With Potentially Clinically Significant Laboratory Findings
Description: Number of patients with potentially clinically significant abnormalities. Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: Up to week 8.
Population: Only participants included in the treated set (TRS) and with non-missing values for each laboratory parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 167 | 171
Participants
  Haematocrit Decrease: number analyzed (Participants) | 167 | 159
  Haematocrit Decrease | 0 | 1
  Haenatocrit Increase: number analyzed (Participants) | 167 | 159
  Haenatocrit Increase | 0 | 0
  Red blood cell ct. Decrease: number analyzed (Participants) | 156 | 160
  Red blood cell ct. Decrease | 0 | 1
  Red blood cell ct. Increase: number analyzed (Participants) | 156 | 160
  Red blood cell ct. Increase | 0 | 0
  MCV Decrease | 0 | 0
  MCV Increase | 0 | 1
  MCHC Decrease: number analyzed (Participants) | 156 | 171
  MCHC Decrease | 0 | 0
  MCHC Increase: number analyzed (Participants) | 167 | 160
  MCHC Increase | 0 | 0
  White blood cell ct. Decrease: number analyzed (Participants) | 156 | 160
  White blood cell ct. Decrease | 1 | 2
  White blood cell ct. Increase: number analyzed (Participants) | 156 | 171
  White blood cell ct. Increase | 0 | 0
  Platelets Decrease: number analyzed (Participants) | 156 | 158
  Platelets Decrease | 0 | 0
  Platelets Increase: number analyzed (Participants) | 156 | 158
  Platelets Increase | 0 | 0
  Eosinophils Decrease: number analyzed (Participants) | 156 | 160
  Eosinophils Decrease | 0 | 0
  Eosinophils Increase: number analyzed (Participants) | 156 | 160
  Eosinophils Increase | 0 | 0
  Basophils Decrease: number analyzed (Participants) | 156 | 160
  Basophils Decrease | 0 | 0
  Basophils Increase: number analyzed (Participants) | 156 | 160
  Basophils Increase | 0 | 0
  Lymphocytes Decrease: number analyzed (Participants) | 156 | 160
  Lymphocytes Decrease | 0 | 0
  Lymphocytes Increase: number analyzed (Participants) | 156 | 160
  Lymphocytes Increase | 0 | 0
  Monocytes Decrease: number analyzed (Participants) | 156 | 160
  Monocytes Decrease | 0 | 0
  Monocytes Increase: number analyzed (Participants) | 156 | 160
  Monocytes Increase | 0 | 0
  Neut., bands (stabs) Decrease: number analyzed (Participants) | 156 | 160
  Neut., bands (stabs) Decrease | 0 | 0
  Neut., bands (stabs) Increase: number analyzed (Participants) | 156 | 160
  Neut., bands (stabs) Increase | 0 | 0
  Sodium Decrease: number analyzed (Participants) | 160 | 163
  Sodium Decrease | 1 | 0
  Sodium Increase: number analyzed (Participants) | 160 | 163
  Sodium Increase | 0 | 0
  Potassium Decrease: number analyzed (Participants) | 159 | 163
  Potassium Decrease | 0 | 0
  Potassium Increase: number analyzed (Participants) | 159 | 163
  Potassium Increase | 0 | 1
  Calcium Decrease: number analyzed (Participants) | 160 | 163
  Calcium Decrease | 0 | 0
  Calcium Increase: number analyzed (Participants) | 160 | 163
  Calcium Increase | 0 | 0
  Chloride Decrease: number analyzed (Participants) | 160 | 163
  Chloride Decrease | 0 | 0
  Chloride Increase: number analyzed (Participants) | 160 | 163
  Chloride Increase | 0 | 0
  Phosphate Decrease: number analyzed (Participants) | 159 | 163
  Phosphate Decrease | 0 | 0
  Phosphate Increase: number analyzed (Participants) | 159 | 163
  Phosphate Increase | 0 | 0
  Bicarbonate Decrease: number analyzed (Participants) | 158 | 161
  Bicarbonate Decrease | 0 | 0
  Bicarbonate Increase: number analyzed (Participants) | 158 | 161
  Bicarbonate Increase | 0 | 0
  AST/GOT, SGOT Decrease: number analyzed (Participants) | 158 | 161
  AST/GOT, SGOT Decrease | 0 | 0
  AST/GOT, SGOT Increase: number analyzed (Participants) | 158 | 161
  AST/GOT, SGOT Increase | 2 | 0
  ALT/GPT, SGPT Decrease: number analyzed (Participants) | 159 | 161
  ALT/GPT, SGPT Decrease | 0 | 0
  ALT/GPT, SGPT Increase: number analyzed (Participants) | 159 | 161
  ALT/GPT, SGPT Increase | 3 | 1
  Alkaline phosphatase Decrease | 0 | 0
  Alkaline phosphatase Increase | 0 | 1
  GGT Decrease: number analyzed (Participants) | 161 | 163
  GGT Decrease | 0 | 0
  GGT Increase: number analyzed (Participants) | 161 | 163
  GGT Increase | 2 | 0
  Creatine kinase Decrease: number analyzed (Participants) | 159 | 161
  Creatine kinase Decrease | 0 | 0
  Creatine kinase Increase: number analyzed (Participants) | 159 | 161
  Creatine kinase Increase | 6 | 3

26. Secondary Outcome: Number of Patients Withdrawn Due to Adverse Events
Description: Number of patients withdrawn due to adverse events.
  Results are reported by treatment regimen (60 mg duloxetine vs. 120 mg duloxetine).
Time Frame: From start of treatment until 3 days after end of treatment, up to 120 days.
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
Number analyzed (Participants) | 167 | 171
Participants | 11 | 9

ADVERSE EVENTS:
Time Frame: From first drug administration until last drug administration (average duration of 55.1 days), plus 3 days, up to 120 days.
Description: Treated Set (TRS): All randomised patients treated with at least one dose of duloxetine. Participants randomised but not treated with at least one dose of duloxetine were excluded, as they cannot contribute information on the drug effect. Adverse Event were analyzed by treatment arm (60 mg vs 120 mg) as prespecified in the statistical analysis plan.
Arm/Group | 60 mg Duloxetine | 120 mg Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/171
Serious Adverse Events (participants affected / at risk) | 6/167 | 6/171
Other Adverse Events (participants affected / at risk) | 67/167 | 54/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 60 mg Duloxetine (N=167) | 120 mg Duloxetine (N=171)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Suicide attempt (Psychiatric disorders) | 4 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 2
Serotonin syndrome (Nervous system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 60 mg Duloxetine (N=167) | 120 mg Duloxetine (N=171)
Nasopharyngitis (Infections and infestations) | 4 | 9
Nausea (Gastrointestinal disorders) | 37 | 21
Constipation (Gastrointestinal disorders) | 8 | 16
Headache (Nervous system disorders) | 26 | 19
Dry mouth (Gastrointestinal disorders) | 9 | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.